CLINICAL TRIAL: NCT05093036
Title: The EZI-PrEP Study: E-Health for Zero Infections - Facilitating Access to and Use of HIV Pre-Exposure Prophylaxis (PrEP) in the Netherlands
Brief Title: E-Health for Zero Infections - Facilitating Access to and Use of HIV Pre-Exposure Prophylaxis (PrEP) in the Netherlands
Acronym: EZI-PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Service of Amsterdam (Other Government)
Collaborators: Public Health Service Rotterdam-Rijnmond (Unknown); Public Health Service Haaglanden (Unknown); Public Health Service Gelderland-Zuid (Unknown); The National Institute for STI and Aids Control in the Netherlands (Soa Aids Nederland) (Unknown); Stichting Aidsfonds (Unknown); DC Pharmacy of DC Klinieken (Unknown)
Responsible Party: Principal Investigator, Dr. Udi Davidovich, Senior researcher (PhD), Public Health Service of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NL74494.018.20
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: Pre-Exposure Prophylaxis (PrEP); Prevention; E-Health
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: We will implement a multi-center, four-arm, non-inferiority randomised controlled trial to evaluate online PrEP care and/or a reduced schedule of monitoring visits against routine (face-to-face) PrEP care at the Centers of Sexual Health (CSH) of the Public Health Services (PHS) (standard-of-care). After eligibility screening and assessment, study participants are randomized (1:1:1:1) to the standard-of-care arm (i.e. location: CSH; 4 annual monitoring visits) or one of three interventions arms: arm 2 (location: CSH; 2 annual monitoring visit), arm 3 (location: online; 4 annual monitoring visits), arm 4 (location: online; 2 annual monitoring visits). In the randomization process, participants will be stratified based on PrEP experience (PrEP-naïve or experienced) and PHS catchment area (4 regions). In each arm, we aim to include at least 25% PrEP-naïve participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: routine PrEP care at the CSH, monitoring 4 times per year (standard-of-care) (No Intervention): Study participants in arm 1 follow routine care procedures, i.e. the number of monitoring visits is four times a year.
  * Experienced PrEP users: first monitoring visit is three months after the enrolment into the study.
  * PrEP-naïve participants: first monitoring visit is one month after enrolment in the study and start of PrEP use. The second monitoring visit is 2 months after the first monitoring contact (3 months after enrolment).
- Arm 2: routine PrEP care at the CSH, monitoring 2 times per year (Experimental): Study participants in arm 2 follow routine care procedures but with a reduced frequency of monitoring visits, i.e. the number of monitoring visits is reduced from four to two times a year. Timing of the first monitoring visit differs per PrEP user type:
  * Experienced PrEP users: first monitoring visit is six months after the enrolment into the study.
  * PrEP-naïve participants: first monitoring visit is one month after enrolment in the study and start of PrEP use. The second monitoring visit is five months after the first monitoring visit (6 months after enrolment).
  Interventions: Other: Variations in PrEP care delivery at public health services
- Arm 3: online PrEP care, monitoring 4 times per year (Experimental): Study participants in arm 3 receive internet-based PrEP care, i.e. video consultations and online-mediated testing for HIV, STIs and renal function, online PrEP ordering and (at home) delivery of PrEP. Monitoring occurs four times per year.
  * Experienced PrEP users: first monitoring contact is three months after the enrolment into the study.
  * PrEP-naïve participants: first monitoring contact is one month after enrolment in the study and start of PrEP use. The second monitoring visit is 2 months after the first monitoring contact (3 months after enrolment).
  Interventions: Other: Variations in PrEP care delivery at public health services
- Arm 4: online PrEP care, monitoring 2 times per year (Experimental): Study participants in arm 4 receive internet-based PrEP care, i.e. video consultations and online-mediated testing for HIV, STIs and renal function, online PrEP ordering and (at home) delivery of PrEP. Monitoring occurs two times per year.
  * Experienced PrEP users: first monitoring contact is six months after the enrolment into the study.
  * PrEP-naïve participants: first monitoring contact is one month after enrolment in the study and start of PrEP use. The second monitoring visit is five months after the first monitoring contact (6 months after enrolment).
  Interventions: Other: Variations in PrEP care delivery at public health services

INTERVENTIONS:
Other: Variations in PrEP care delivery at public health services — Variations on routine PrEP care at the Public Health Services in the Netherlands: online PrEP care and reduced frequency of monitoring
  Arms: Arm 2: routine PrEP care at the CSH, monitoring 2 times per year; Arm 3: online PrEP care, monitoring 4 times per year; Arm 4: online PrEP care, monitoring 2 times per year

SUMMARY:
Offering PrEP care online and reducing the frequency of monitoring may increase access to HIV PrEP. The objective of this study is to assess the non-inferiority of an internet-based HIV PrEP-service and reduced frequency of monitoring visits in comparison to standard-of-care at the Public Health Service in 4 regions in the Netherlands: Amsterdam, Rotterdam-Rijnmond, Haagland and Gelderland-Zuid.

DETAILED DESCRIPTION:
Rationale: The population impact of HIV pre-exposure prophylaxis (PrEP) largely depends on the uptake and consistent use of PrEP by people at high risk for HIV infection. In the Dutch National PrEP Programme (NPP), PrEP care consists of quarterly monitoring visits, which includes testing for HIV, sexually transmitted infections (STIs) and renal function, and provision of combination tablets of tenofovir disoproxil fumarate and emtricitabine. PrEP care is available for men who have sex with men (MSM) and transgender persons (TGP) at low cost through the centers for sexual health (CSH) of public health services (GGD's). Offering PrEP care online and reducing the frequency of monitoring may increase access to PrEP.

Objective: To assess the non-inferiority of an internet-based HIV PrEP-service and reduced frequency of monitoring visits in comparison to standard-of-care at the Public Health Service.

Study design: Randomised, non-blinded, controlled, parallel group, non-inferiority trial.

Study population: MSM and TGP of 18 years of age or older who are eligible for HIV PrEP according to NPP guidelines based on self-reported sexual behavior indicating HIV risk.

Intervention: The study takes place in four GGD regions in the Netherlands: Amsterdam, Haaglanden, Rotterdam-Rijnmond and Gelderland-Zuid. Participants will be assigned to one of four arms: (1) routine care with quarterly monitoring at CSH; (2) routine care with biannual monitoring at CSH; (3) internet-based PrEP-care (i.e. video consultations and online-mediated testing for HIV, STIs and renal function) with quarterly monitoring; (4) internet-based PrEP-care with biannual monitoring. Each participant will be followed for 18 months.

Main study parameters/endpoints: The primary outcome is adherence to PrEP, determined by self-reported daily data on pill-intake and sexual behavior. Non-adherence is defined as a PrEP-less and condom-less anal sex act with a casual partner. Secondary outcomes include the incidence of HIV and Hepatitis C virus infections and bacterial STIs; creatinine clearance, glycosuria and proteinuria; retention in PrEP-care; psychosocial health; and acceptance and usability of the internet-based PrEP service.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Meeting the eligibility criteria of the NPP i.e. being a MSM or transgender persons who in the 6 months prior to the PrEP-request/PrEP-consultation:

  * Had anal sexual intercourse without a condom with a male partner with an un-known HIV status, and/or;
  * Had anal sexual intercourse without a condom with a male partner with a known HIV-positive status and a detectable viral load, and/or;
  * Was diagnosed with a rectal STI, and/or;
  * Received a prescription for post-exposure prophylaxes (PEP);
* Living in the catchment area of one of the participating GGD regions;
* Having a smartphone, internet access and email address;
* Sufficient understanding of Dutch or English; and
* Signed informed consent.

Exclusion Criteria:

* HIV infection;
* Chronic or acute Hepatitis B virus infection;
* Diminishing renal function:
* eGFR less than 60 mL/min/1.73m2;
* Other renal problems, as diagnosed by a physician and advised against using TFV;
* Chronic use of medication that interacts with TFV/FTC e.g. NSAIDs.
* Other medical conditions that require special attention when using PrEP, such as osteoporosis or other bone diseases;
* Unlikely, in the opinion of the clinician, to comply with the study requirements or procedures;
* Participating in another study that affects the primary or secondary outcome measures of our study;
* Investigators or otherwise dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to PrEP regimen | 18 months for each individual study participant
  Non-adherence is defined as a PrEP-less and condom-less anal sex act with a casual partner, termed an unprotected act (UA). Self-reported daily data on sexual behaviour, pill intake and condom use are recorded in an electronic diary. Using these data, we will count the number of UAs (n), and the person-months at risk (pmar) per person; this will yield the incidence rate (IR) per person month (= n / pmar). This will be done for each study arm separately.

CONTACTS AND LOCATIONS:
Overall Officials: Udi Davidovich, PhD, Principal Investigator — Public Health Service of Amsterdam; Maarten Schim van der Loeff, Principal Investigator — Public Health Service of Amsterdam
Locations (4):
- Netherlands (4):
  - Public Health Service of Amsterdam, Amsterdam
  - Public Health Service Gelderland-Zuid, Nijmegen
  - Public Health Service Rotterdam-Rijnmond, Rotterdam
  - Public Health Service Haaglanden, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groot Bruinderink ML, Boyd A, Coyer L, Boers S, Blitz L, Brand JM, Gotz HM, Stip M, Woudstra J, Yap K, Vermey K, Matser A, Feddes AR, Jongen VW, Prins M, Hoornenborg E, van Harreveld F, Schim van der Loeff MF, Davidovich U. Online-Mediated HIV Pre-exposure Prophylaxis Care and Reduced Monitoring Frequency for Men Who Have Sex With Men: Protocol for a Randomized Controlled Noninferiority Trial (EZI-PrEP Study). JMIR Res Protoc. 2023 Nov 8;12:e51023. doi: 10.2196/51023. PMID 37938875